CLINICAL TRIAL: NCT04584554
Title: Enhancing the Transition From Hospital to Home for Patients With Traumatic Brain Injury and Families
Acronym: R03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00103181
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Brain Injuries, Traumatic; Transitional Care; Family Members; Patients
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: 15 patient/family dyads will undergo intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: BETTER Transitional Care Intervention

INTERVENTIONS:
Behavioral: BETTER Transitional Care Intervention — Patient and family will receive pre- and post-discharge support and education from interventionist.

SUMMARY:
Despite high risks of readmission and complex medical needs, there are no transitional care standards in the U.S. for patients with moderate-to-severe traumatic brain injury (TBI) discharged home from acute hospital care without inpatient rehabilitation. To enhance the standard of TBI care, we will develop and refine a patient- and family-centered TBI transitional care intervention that addresses specific needs and preferences for patients with TBI (age < 65 years) and families and will assess the feasibility, acceptability, and preliminary efficacy of the intervention.

DETAILED DESCRIPTION:
Despite high risks of readmission and complex medical needs, there are no transitional care standards in the U.S. for patients with moderate-to-severe traumatic brain injury (TBI). Patients with moderate-to-severe TBI (age < 65 years) discharged home from acute hospital care without inpatient rehabilitation have cognitive, physical, behavioral, and emotional impairments that affect their abilities to independently self-manage their health, wellness, and activities of daily living. Activity limitations often result in increased family involvement for managing the person's care. The complexity of needs combined with the fragmentation of healthcare services creates the perfect storm for mismanaged symptoms, adverse health events, readmissions, and a lower likelihood of return to work and school. Transitional care is defined as actions in the clinical encounter designed to ensure the coordination and continuity of healthcare for patients transferring between different locations or levels of care in close geographic proximity. In other patient groups who experience acute events (e.g., stroke, myocardial infarction), transitional care management has led to improved patient and family outcomes. Although preliminary research shows that patients with TBI and families desire and could benefit from interventions to support the transition from acute hospital care to home, the strength of evidence on this topic is low. TBI transitional care interventions developed to date are ineffective in improving functional outcomes and do not incorporate family needs. Thus, the purpose of our study is to first develop and refine a patient- and family-centered TBI transitional care intervention to support patients with moderate-to-severe TBI and their family caregivers during the transition home from acute hospital care. The intervention will aim to improve quality of life for patients with TBI, reduce strain for their family caregivers, and direct patients and families to appropriate resources and care that is concordant with their health-related goals. Second, we will examine the feasibility and acceptability and assess the preliminary efficacy of the TBI transitional care intervention. The primary outcome will be patient quality of life at 16 weeks post-discharge. This study will also examine secondary outcomes at 16 weeks post-discharge, including family caregiver strain and preparedness for the caregiving role, and patient and family caregiver self-efficacy and healthcare utilization. The new knowledge generated from the proposed research will guide the research team in designing and conducting an NIH R01 implementation-effectiveness clinical trial of the TBI transitional care intervention and will ultimately enhance the standard of care for patients with TBI discharged home from acute hospital care and families

ELIGIBILITY:
Inclusion Criteria:

* Patients: age 18-64 years, diagnosis of mild-moderate TBI based on Glasgow Coma Scale score of 9-14; sufficient cognitive functioning and oral communication skills to participate (as determined by Galveston Orientation and Amnesia Test); set to be discharged directly home from acute hospital care; and has smart phone or computer with internet access.
* Family caregiver: age 18 years or older, primary caregiver for patient post-discharge (i.e., plans to live in same home as person or have direct contact with person >10 hours/week); and has smart phone or computer with internet access.

Exclusion Criteria:

* Patients: who do not have a family caregiver who is willing to participate; prior neurological disorder affecting the brain or language or learning disability

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tolu O Oyesanya, PhD, RN, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Please contact PI for underlying research materials.

REFERENCES:
- [Derived] Oyesanya TO, Loflin C, You H, Kandel M, Johnson K, Strauman T, Yang Q, Hawes J, Byom L, Gonzalez-Guarda R, Van Houtven C, Agarwal S, Bettger JP. Design, methods, and baseline characteristics of the Brain Injury Education, Training, and Therapy to Enhance Recovery (BETTER) feasibility study: a transitional care intervention for younger adult patients with traumatic brain injury and caregivers. Curr Med Res Opin. 2022 May;38(5):697-710. doi: 10.1080/03007995.2022.2043657. Epub 2022 Mar 2. PMID 35174756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trained research coordinators screened the electronic medical record daily to determine eligible patients. TCMs recruited the patient/family dyads. First, the TCM contacted eligible patients by phone 24-72 hours before discharge to determine interest in participating and obtain additional eligibility information. Interested and eligible patients were asked to identify the caregiver they preferred to participate with them and to share the caregiver's name and contact information.
Pre-assignment Details: 15 patient-caregiver dyads started the study.
Groups:
- Intervention Patient-Caregiver Dyad - Patient; Intervention Patient-Caregiver Dyad - Caregiver: BETTER Transitional Care Intervention: Patient and family will receive pre- and post-discharge support and education from interventionist.
Period: Overall Study
Arm/Group | Intervention Patient-Caregiver Dyad - Patient | Intervention Patient-Caregiver Dyad - Caregiver
Started | 15 | 16
Completed | 13 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Patient-Caregiver Dyad - Patient: BETTER Transitional Care Intervention: Patient will receive pre- and post-discharge support and education from interventionist.
- Intervention Patient-Caregiver Dyad - Family Caregivers: BETTER Transitional Care Intervention: Family will receive pre- and post-discharge support and education from interventionist.
- Total: Total of all reporting groups
Arm/Group | Intervention Patient-Caregiver Dyad - Patient | Intervention Patient-Caregiver Dyad - Family Caregivers | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.07 (15.15) | 43.38 (10.45) | 41.25 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life as Measured by the Short Form-36 (SF-36)
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scores on each item are summed and averaged (range: 0=worst to 100=best).
Time Frame: Baseline (24-72 hours pre-discharge) and 16-weeks post-discharge
Population: Younger adults (age 18-64) with mild, moderate, or severe TBI discharged home from acute hospital care without inpatient rehabilitation. Not collected on caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Patient-Caregiver Dyad - Patient
Number analyzed (Participants) | 15
score on a scale | 47.97 (24.93)

2. Secondary Outcome: Change in Preparedness for Caregiving Scale (CPS)
Description: The CPS is a caregiver self-rated instrument that consists of eight items that asks caregivers how well prepared they believe they are for multiple domains of caregiving. Responses are rated on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). Total score range is 0 to 32, where a higher score indicates the caregiver feels more prepared for caregiving.
Time Frame: Baseline (24-72 hours pre-discharge) and 16-weeks post-discharge
Population: Family caregivers of patients with TBI. Not collected on patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Patient-Caregiver Dyad - Caregiver
Number analyzed (Participants) | 16
score on a scale | 25.75 (8.02)

3. Other Pre Specified Outcome: Change in Health Service Utilization Inventory
Description: Health service utilization
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Modified Caregiver Strain Index
Description: Caregiver strain
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Self-efficacy for Managing Chronic Conditions
Description: Self-efficacy
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

6. Post Hoc Outcome: Change in PART-O
Description: Participation
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

7. Post Hoc Outcome: Change in Glasgow Outcome Scale-Extended
Description: Global Outcome
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

8. Post Hoc Outcome: Change in PTSD Checklist
Description: Psychiatric Status (PTSD)
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

9. Post Hoc Outcome: Change in Interpersonal Processes of Care
Description: Perceived Discrimination in Health Settings
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

10. Post Hoc Outcome: Change in Satisfaction With Life
Description: Satisfaction With Life
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

11. Post Hoc Outcome: Change in Rivermead Post Concussion Questionnaire
Description: TBI Symptoms
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

12. Post Hoc Outcome: NeuroQOL Measures (Short Form)
Description: Functional and cognitive status
Time Frame: 16 weeks post-discharge
Reporting Status: Not Posted

13. Post Hoc Outcome: Change in Patient Health Questionnaire (PHQ-9)
Description: Psychiatric status
Time Frame: Baseline (24-72 hours pre-discharge) and 8- and 16-weeks post-discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 weeks post-discharge
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04584554/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04584554/ICF_001.pdf